CLINICAL TRIAL: NCT00240643
Title: A Randomized, Double Blind, Double Dummy, Parallel Group, Placebo Controlled Study to Evaluate the Pharmacodynamic and Pharmacokinetic Response and Safety and Tolerability of SB424323 (250mg, 375mg and 500 mg) Administered Twice Daily for 16 Weeks, on Top of Asprin (325mg, qd) in Men and Women With Non Valvular Atrial Fibrillation at a Low or Intermediate Risk for Stroke
Brief Title: Use Of SB424323 With Aspirin In Non-Valvular Atrial Fibrillation In Patients At A Low Or Intermediate Risk For Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Cheri Hudson; Clinical Disclosure Advisor, GSK Clinical Disclosure
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 101724
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Fibrillation, Atrial; Atrial Fibrillation
Keywords: non valvular atrial fibrillation; stroke; aspirin
MeSH Terms: conditions — Atrial Fibrillation; Stroke

INTERVENTIONS:
Drug: SB424323

SUMMARY:
This study will allow determination of the pharmacokinetic and pharmacodynamics of SB424323 in a relevant population. The data from this study will be used along with other data to aid in choosing the most appropriate dose for the later phase study.

DETAILED DESCRIPTION:
A randomized, double blind, double dummy, parallel group, placebo controlled study to evaluate the pharmacodynamic and pharmacokinetic response and safety and tolerability of SB424323 (250 mg, 375 mg and 500 mg) administered twice daily for 16 weeks, on top of aspirin (325 mg, qd) in men and women with non valvular atrial fibrillation at a low or intermediate risk for stroke

ELIGIBILITY:
Inclusion Criteria:

* Patients with non valvular atrial fibrillation and any of the following:
* </= 60 years old with no heart disease.
* 60 years old with heart disease but no risk factors.
* >/=60 years old and </=75 years old with no risk factors and no heart disease.
* Must be able to take aspirin.

Exclusion Criteria:

* Previous heart attack or stroke.
* History of high blood pressure, diabetes or a prior blood clot.
* Liver or kidney disease.
* Need for anti-thrombotic or anti-platelet drugs.
* Need for cardiovascular medicines.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Actual)
Dates: Start 2005-11; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Relationship between anti IIa (a biomarker)and the dose of SB424323.

SECONDARY OUTCOMES:
Blood levels of SB424323 during the study. Number of strokes, transient ischemic attacks or systemic embolism during the study. Changes in laboratory tests during the study.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (101):
- United States (9):
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Troy, Michigan
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Camp Hill, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Walla Walla, Washington
  - GSK Investigational Site, Milwaukee, Wisconsin
- Argentina (7):
  - GSK Investigational Site, Buenos Aires, Buenos Aires
  - GSK Investigational Site, Capital Federal, Buenos Aires
  - GSK Investigational Site, Capital Fefderal, Buenos Aires
  - GSK Investigational Site, Córdoba, Córdoba Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Moron-Provincia de Buenos Aires
- Belgium (2):
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Linkebeek
- Brazil (2):
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, São Paulo, São Paulo
- Canada (12):
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Burlington, Ontario
  - GSK Investigational Site, Grimsby, Ontario
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Newmarket, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Greenfield Park, Quebec
  - GSK Investigational Site, Longueuil, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Saint-Lambert, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec
- Denmark (2):
  - GSK Investigational Site, Aarhus
  - GSK Investigational Site, Frederiksberg
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- France (4):
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Mont-de-Marsan
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Tours
- Germany (13):
  - GSK Investigational Site, Künzing, Bavaria
  - GSK Investigational Site, Northeim, Lower Saxony
  - GSK Investigational Site, Weyhe-Leeste, Lower Saxony
  - GSK Investigational Site, Chemnitz, Saxony
  - GSK Investigational Site, Ebersbach, Saxony
  - GSK Investigational Site, Königsbrück, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Leisnig, Saxony
  - GSK Investigational Site, Markkleeberg, Saxony
  - GSK Investigational Site, Wolmirstedt, Saxony-Anhalt
  - GSK Investigational Site, Bad Segeberg, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
  - GSK Investigational Site, Jena, Thuringia
- GSK Investigational Site, Athens, Greece
- Hungary (3):
  - GSK Investigational Site, Sopron
  - GSK Investigational Site, Székesfehérvár
  - GSK Investigational Site, Szolnok
- India (4):
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Hyderabad
  - GSK Investigational Site, Mumbai
  - GSK Investigational Site, New Delhi
- Italy (4):
  - GSK Investigational Site, Catanzaro, Calabria
  - GSK Investigational Site, Caserta, Campania
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Città Della Pieve (PG), Umbria
- GSK Investigational Site, Riga, Latvia
- GSK Investigational Site, México, Mexico
- Netherlands (3):
  - GSK Investigational Site, Delft
  - GSK Investigational Site, The Hague
  - GSK Investigational Site, Utrecht
- New Zealand (4):
  - GSK Investigational Site, Auckland
  - GSK Investigational Site, Christchurch
  - GSK Investigational Site, Hamilton
  - GSK Investigational Site, Takapuna, Auckland
- Norway (3):
  - GSK Investigational Site, Elverum
  - GSK Investigational Site, Oslo
  - GSK Investigational Site, Skien
- Romania (2):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Târgu Mureş
- South Korea (2):
  - GSK Investigational Site, Kwangju
  - GSK Investigational Site, Seoul
- Spain (6):
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Cadiz
  - GSK Investigational Site, Leganés
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Sant Joan d'Alacant
- Sweden (3):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Uppsala
- GSK Investigational Site, Taipei, Taiwan
- Thailand (2):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai
- United Kingdom (8):
  - GSK Investigational Site, Glasgow, Lanarkshire
  - GSK Investigational Site, Harrow, Middlesex
  - GSK Investigational Site, Northwood, Middlesex
  - GSK Investigational Site, Birmingham, West Midlands
  - GSK Investigational Site, Antrim
  - GSK Investigational Site, Dundee
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, York